CLINICAL TRIAL: NCT07093463
Title: The Benefit of Colon-delivered Riboflavin (Riboflavin-cd) vs. Conventional Riboflavin on Gut Microbiota Composition and Metabolic Output in Healthy Aging Subjects - a Pilot Proof of Concept Study
Brief Title: Colon-delivered Riboflavin and Gut Microbiota Composition
Acronym: CONCOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Collaborators: Analyze & Realize (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DSM/230702; DSM/011224 (Other: Cro)
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Microbiome Dysbiosis; Gut Health
Keywords: elderly; microbiome; colon delivered b-vitamins; riboflavin
MeSH Terms: interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Colon-delivered riboflavin (Active Comparator): This arm includes 10 mg of colon-delivered riboflavin
  Interventions: Dietary Supplement: Colon-delivered riboflavin
- Conventional riboflavin (Active Comparator): This arm includes 10 mg of conventional riboflavin that will be absorbed in the upper small intestine and not reach the colon
  Interventions: Dietary Supplement: Conventional riboflavin
- Placebo (Placebo Comparator): This arm includes 10 mg of microcrystalline cellulose
  Interventions: Other: Microcrystalline Cellulose

INTERVENTIONS:
Dietary Supplement: Colon-delivered riboflavin — 10 mg of colon-delivered riboflavin
  Arms: Colon-delivered riboflavin
Dietary Supplement: Conventional riboflavin — 10 mg of conventional riboflavin
  Arms: Conventional riboflavin
Other: Microcrystalline Cellulose — 10 mg microcrystalline cellulose
  Arms: Placebo

SUMMARY:
Recent studies suggest B-vitamins such as riboflavin to possess prebiotic-like effects. However, there is still a lack of understanding of the exact host health benefits vs. conventional systemically available vitamin forms. The present study explores the benefit of colon-delivered vitamin B2 vs. conventional vitamin B2 in comparison to placebo in an aging population on gut microbiota and metabolic activity as well as gut health.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals providing written informed consent for participation in the study and data processing
2. Female and males between 50 and 70 years of age
3. For females only: Menopausal as marked by at least 1 year since the last menstrual bleeding
4. Individuals with a BMI between 18.5 - 29.9 Kg/m2
5. Individuals with stable body weight (≤5% change) over the past 3 months prior to V1
6. Individuals with self-reported moderate bowel complaints in at least last 3 months prior to V1
7. Individuals with GSRS score suggestive of moderate bowel complaints, as assessed at V1, for the average condition over the 4 last weeks (all GSRS items have to be answered at V1): • indigestion score 3-5 or constipation score 3-5 or diarrhoea score 3-5
8. Individuals with a general good health, as determined by questioning, clinical examination and vital signs (blood pressure, pulse rate) by the investigator at V1
9. Individuals willing to avoid consuming gut microbiome modulating dietary supplements, prebiotic, probiotic, synbiotic or fibre-rich supplements during the entire study duration
10. Individuals willing to maintain current level of physical activity throughout the entire study duration
11. If individuals are taking chronic medications (e.g., antihypertensive medications), they must be willing and expected to maintain the same dosage throughout the study

Exclusion Criteria:

1. Individuals who are hypersensitive/intolerant to any of the components of the Investigational product or the standardised diet addition (inulin)
2. Individuals who have taken systemic antibiotics within the previous 3 months prior to Baseline (V2) or are expected to be taking any during the study
3. Individuals who consumed microbiome modulating dietary supplements, prebiotic, probiotic, or fibre-rich supplements within 4 weeks prior to the baseline (V2)
4. Individuals who are currently regularly using systemic steroids, proton pump inhibitors, H2 blocker, antacids (however, sporadic use during the study if needed is allowed, but not within 8 hours before each visit), metformin if started less than 6 months prior to V1, or immunosuppressant medication.
5. Individuals who have a history of drug abuse in the previous 5 years and/or alcohol abuse at the time of enrolment (>11 units/week for women; >17 units/week for men; unit: approx. 125 mL of wine or similar / approx. 30 mL of spirits

   / approx. 280 mL beer or similar); Is currently in treatment for alcohol/substance abuse; Has been diagnosed with alcohol/substance abuse disorder)
6. Individuals who are a smoker or vaper
7. Individuals who are vegetarian or vegan
8. Individuals who have made any major dietary changes in the past 3 months prior to Baseline (V2)
9. Individuals who have planned major changes in the lifestyle (i.e., diet, dieting, exercise level, significant travel) during the duration of the study.
10. Individuals who have a currently present active eating disorder
11. Individuals with self-reported food allergy / intolerance (e.g., lactose, gluten, fructose), as determined by the study investigator
12. Clinical significance for any of screening laboratory test results from the blood draw at V1, as per investigator's judgement
13. Individuals with a self-reported fibre-rich regular diet, as per investigator's judgement
14. Individuals who have a (self-reported) gastrointestinal disorder/disease (e.g., chronic/recurrent diarrhoea, inflammatory bowel disorder, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers, bile acid malabsorption) or previous gastrointestinal surgery (such as bariatric surgery, colon specific surgical interventions etc.), which in the opinion of the investigator would impact the study outcomes
15. Individuals with GSRS assessed at V1 for the average condition over the 4 last weeks prior to V1 for any score (abdominal pain, reflux score, indigestion, constipation, diarrhoea) >5 (all GSRS items have to be answered at V1)
16. Individuals who have severe or uncontrolled conditions such as type 2 diabetes (FBG ≥ 150 mg/dl from blood draw at V1), psychiatric disorder, respiratory or cardiac illness or any other condition which in the opinion of the investigator would impact the study outcomes
17. Individuals who have a history of any gastrointestinal cancer
18. Individuals who are severely immunocompromised
19. Individuals with alarm features in the past 3 months prior to V1 such as unintentional weight loss (≤5% change), fever, anorectal problems, blood in stool, vomiting
20. Individuals who, in the opinion of the investigator are considered to be poor attendees or unlikely for any reason to be able to comply with the study requirements
21. If Individuals have been in a recent experimental study, this must have been completed not less than 30 days prior to this study

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Microbial alpha diversity | 4 weeks' daily consumption of 10 mg of colon delivered riboflavin (riboflavin-cd)
  Variation D28 - D0 in the faecal microbial alpha diversity (Observed richness, Inverse Simpson index, Shannon index)

SECONDARY OUTCOMES:
Microbial alpha diversity | 8 weeks' daily consumption of 10 mg of colon delivered riboflavin (riboflavin-cd) including 5 g of dietary fiber inulin per day as a standardised addition to the subjects daily diet from week 4 to week 8.
  Variation D56 - D0 in the faecal microbial alpha diversity (Observed richness, Inverse Simpson index, Shannon index)
Microbial composition | 8 weeks' daily consumption of 10 mg of colon delivered riboflavin (riboflavin-cd) including 5 g of dietary fiber inulin per day as a standardised addition to the subjects daily diet from week 4 to week 8.
  Variations D28 - D0 and D56 - D0 in faecal microbial composition, assessed in terms of relative abundance of components at phylum, family, genus and species level and beta diversity (including Jaccard and Bray- Curtis dissimilarity indices)
Faecal organic acid | 8 weeks' daily consumption of 10 mg of colon delivered riboflavin (riboflavin-cd) including 5 g of dietary fiber inulin per day as a standardised addition to the subjects daily diet from week 4 to week 8.
  Variations D28 - D0 and D56 - D0 in faecal organic acid levels (acetate, propionate, butyrate, valerate, lactate)
Faecal riboflavin | 8 weeks' daily consumption of 10 mg of colon delivered riboflavin (riboflavin-cd) including 5 g of dietary fiber inulin per day as a standardised addition to the subjects daily diet from week 4 to week 8.
  Variations D28 - D0 and D56 - D0 in faecal concentrations of riboflavin
Fecal redox potential | 8 weeks' daily consumption of 10 mg of colon delivered riboflavin (riboflavin-cd) including 5 g of dietary fiber inulin per day as a standardised addition to the subjects daily diet from week 4 to week 8.
  Variations D28 - D0 and D56 - D0 in fecal redox potential level
fecal pH | 8 weeks' daily consumption of 10 mg of colon delivered riboflavin (riboflavin-cd) including 5 g of dietary fiber inulin per day as a standardised addition to the subjects daily diet from week 4 to week 8.
  Variations D28 - D0 and D56 - D0 in fecal pH
Fecal calprotectin | 8 weeks' daily consumption of 10 mg of colon delivered riboflavin (riboflavin-cd) including 5 g of dietary fiber inulin per day as a standardised addition to the subjects daily diet from week 4 to week 8.
  Variations D28 - D0 and D56 - D0 in fecal calprotectin
Plasma Intestinal barrier markers | 8 weeks' daily consumption of 10 mg of colon delivered riboflavin (riboflavin-cd) including 5 g of dietary fiber inulin per day as a standardised addition to the subjects daily diet from week 4 to week 8.
  Variations D28 - D0 and D56 - D0 in plasma intestinal barrier markers (LBP, I-FABP, zonulin and DAO)
Gastrointestinal complaints | 8 weeks' daily consumption of 10 mg of colon delivered riboflavin (riboflavin-cd) including 5 g of dietary fiber inulin per day as a standardised addition to the subjects daily diet from week 4 to week 8.
  Variations D28 - D0 and D56 - D0 in gastrointestinal complaints assessed by the gastrointestinal Symptom Rating Scale (GSRS) (reflux, abdominal pain, indigestion, diarrhoea, constipation)
Stool consistency and frequency | 8 weeks' daily consumption of 10 mg of colon delivered riboflavin (riboflavin-cd) including 5 g of dietary fiber inulin per day as a standardised addition to the subjects daily diet from week 4 to week 8.
  Variations D28 - D0 and D56 - D0 in stool consistency as assessed by Bristol Stool Form Scale (BSFS) and frequency
Quality of life (Short-Form Health Survey (SF-36)) | 8 weeks' daily consumption of 10 mg of colon delivered riboflavin (riboflavin-cd) including 5 g of dietary fiber inulin per day as a standardised addition to the subjects daily diet from week 4 to week 8.
  Variations D28 - D0 and D56 - D0 in quality of life as assessed by the Short-Form Health Survey (SF-36)
Investigational product (IP) perceived benefit | 8 weeks' daily consumption of 10 mg of colon delivered riboflavin (riboflavin-cd) including 5 g of dietary fiber inulin per day as a standardised addition to the subjects daily diet from week 4 to week 8.
  Variations D28 - D0 and D56 - D0 in Investigational product (IP) perceived benefit assessed by a by a 5 point Likert scale

OTHER OUTCOMES:
Plasma riboflavin concentrations | 8 weeks' daily consumption of 10 mg of colon delivered riboflavin (riboflavin-cd) including 5 g of dietary fiber inulin per day as a standardised addition to the subjects daily diet from week 4 to week 8.
  Variations D28 - D0 and D56 - D0 in Plasma riboflavin concentrations
Plasma immune markers | 8 weeks' daily consumption of 10 mg of colon delivered riboflavin (riboflavin-cd) including 5 g of dietary fiber inulin per day as a standardised addition to the subjects daily diet from week 4 to week 8.
  Variations D28 - D0 and D56 - D0 in plasma immune markers (IL-6, IL-10, TNF alpha)

CONTACTS AND LOCATIONS:
Locations (1):
- analyze & realize GmbH, Berlin, State of Berlin, Germany